CLINICAL TRIAL: NCT06027190
Title: To Investigate the Clinical Efficacy of Optical 3D Navigation Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Achalasia, Optimize the Treatment Parameters, and Provide a Noninvasive Treatment Strategy for Achalasia
Brief Title: Randomized Controlled Study of Optical 3D Navigated Repetitive Transcranial Magnetic Stimulation for Achalasia.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Nina (Other)
Responsible Party: Sponsor-Investigator, Zhang Nina, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-160-02
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Achalasia; Transcranial Magnetic Stimulation, Repetitive; Vagus Nerve Motor Disorder; Functional Magnetic Resonance Imaging
Keywords: Achalasia; rTMS; fMRI; Non-invasive
MeSH Terms: conditions — Esophageal Achalasia; Vagus Nerve Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: In patients with achalasia diagnosed by clinical symptoms, HREM and barium meal examination, functional connectivity analysis of DMV with three brain regions (precentral gyrus, postcentral gyrus and insula) was performed by scanning T1 structural magnetic resonance imaging, and brain regions with the strongest positive functional connectivity with DMV were selected as individualized rTMS targets by optical 3D navigation. All patients were randomly divided into four groups: sham-rTMS group, 5Hz-rTMS group, 10Hz-rTMS group, and 30Hz-rTMS group, and each group received acute and chronic stimulation, respectively.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Sham Comparator): Intervention Name and Specification: Placebo coil (Magstim Company, Whitland, UK): looks and sounds consistent with true coil but does not produce current stimulation.
  Interventions: Device: Sham
- rTMS group (Experimental): 1. 5Hz-rTMS group
  2. 10Hz-rTMS group
  3. 30Hz-rTMS group
  Intervention Name and Specification:
  1. Transcranial magnetic stimulator (M-100 Ultimate, Yingzhi Technology Co., Ltd., China)
  2. 70 mm diameter figure-of-eight coil (BY90A, Yingzhi Technology Co., Ltd., China).
  Each group received acute and chronic stimulation, respectively. In the acute stimulation stage, patients only needed to do rTMS once, and HREM and HRV were administered before and after rTMS; in the chronic stimulation stage, patients received 25 minutes of rTMS true stimulation each time a day for 20 times, which was completed within 30 days, and the true stimulation parameters were the same as those of acute stimulation.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Intervention Name and Specification
  1. Transcranial magnetic stimulator (M-100 Ultimate, Yingzhi Technology Co., Ltd., China) .
  2. 70-mm-diameter figure-of-eight coil (BY90A, Yingzhi Technology Co., Ltd., China). 3) Placebo coil (Magstim Company, Whitland, UK): the appearance and sound were consistent with the true coil, but no current stimulation was produced.
  Arms: rTMS group
Device: Sham — Placebo coil (Magstim Company, Whitland, UK):
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to investigate the clinical efficacy of repetitive transcranial magnetic stimulation in the treatment of achalasia in patients diagnosed with achalasia by comprehensive evaluation of clinical symptoms, HREM, and barium meal examination, optimize rTMS treatment parameters, and provide an effective and noninvasive new treatment strategy for achalasia. The main questions it aims to answer are:

1. To investigate the clinical efficacy of individualized treatment of achalasia with optical 3D navigation repetitive transcranial magnetic stimulation.
2. Optimize rTMS parameters to achieve the best clinical treatment.

Participants will need to fill out the Eckardt score scale and SF-36 quality of life scale, undergo cranial T1 structural magnetic resonance for functional connectivity analysis, and select the brain region with the strongest positive functional connectivity to the DMV as the rTMS target. All patients were randomly divided into four groups: sham-rTMS group, 5Hz-rTMS group, 10Hz-rTMS group, and 30Hz-rTMS group, and each group received acute and chronic stimulation, respectively. In the acute stimulation stage, patients only need to do rTMS once, and HREM and HRV detection are given before and after rTMS (stimulation for 1s, interval for 4s, 10 pulses per second, receiving a total of 3000 pulses); in the chronic stimulation stage, patients receive 25 minutes of rTMS actual stimulation or sham stimulation each time, lasting for 20 times, which is completed within 30 days, and the actual stimulation parameters are the same as those of acute stimulation, and the sham stimulation coil is consistent with the appearance and sound of proper stimulation, but there is no substantial stimulation. High-definition esophageal manometry, timed barium meal, heart rate coefficient of variation, and serum neurotransmitters were performed before and after chronic stimulation. Finally, a weekly telephone follow-up was performed for 12 weeks, including Eckardt score and SF-36 quality of life scale.

DETAILED DESCRIPTION:
Study hypothesis: By analyzing the strongest resting-state functional connectivity between DMV and right precentral gyrus, left postcentral gyrus, and left brain leads in achalasia patients, individualized rTMS treatment with optical 3D navigation was applied to relax LES and relieve the clinical symptoms of dysphagia.

Statistical methods: SPSS 25.0 software was used to process the data, symptom score, manometry parameters, serum transmitters and other quantitative indicators. If they met the normal distribution, they were expressed as Mean ± SD. The t-test was performed for the comparison between the two groups; if they did not obey the normal distribution, the median (quartile) was used for statistical description. The rank sum test was used for the comparison between the two groups. Enumeration data were described using number of cases (percentage), and X2 test, corrected X2 test, or Fisher exact test were performed for comparison between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old, less than 75 years old;
* Clinical symptoms evaluation, HREM, esophageal barium meal examination confirmed the diagnosis of achalasia;
* Willing to sign informed consent.

Exclusion Criteria:

* Presence of metal hardware in close contact with the discharge coil (e.g., cochlear implant, internal pulse generator, or drug pump). Note: Cochlear implants include electrodes, magnets, loop antennas, and electronic chips under the scalp implanted in the cochlea;
* Intracranial metal implants;
* Patients with cardiac pacemakers, vagal nerve stimulation (VNS) systems, spinal cord stimulators, and deep brain stimulation implanted with pulse generators should be used with caution;
* People at higher risk of noisy hearing loss and patients with hypoacusis symptoms should be used with caution;
* Pregnancy;
* Severe or recent heart disease;
* Personal history of epilepsy, use of known drugs that lower the seizure threshold, and other factors that may lower the seizure threshold (e.g., lack of sleep, infection, and alcohol abuse);
* Increased intracranial pressure;
* Acute phase of intracranial infection and hemorrhagic disease;
* Contraindications to MRI examination or claustrophobia;
* Refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Eckardt score | Measured immediately after intervention.
  The Eckardt scoring system is used to assess the severity of symptoms, with 0 to 1 in grade 0, 2 to 3 in grade I., 4 to 6 in grade II., and > 6 in grade III. The more severe the symptoms, the higher the score, and can also be used for efficacy assessment.
Real-time esophageal barium meal examination | Measured immediately after intervention.
  The severity of the patient 's condition and the therapeutic effect were evaluated by defining the height and maximum width of the residual barium area.
High-resolution esophageal manometry（HREM） | Measured immediately after intervention.
  HREM is the gold standard for the diagnosis of achalasia of cardia (AC), which can assess the relaxation ability of the lower esophageal sphincter (LES) and the contraction ability of the esophageal body. HREM dynamically collects the mean pressure data of multiple parts of the whole esophagus in real time, and converts the linear manometry pattern into color pressure topography. The basic manometry parameters include integrated relaxation pressure (IRP) and lower esophageal sphincter pressure (LESP), which can more truly reflect the relaxation function of the gastroesophageal junction (EGJ) and are the key indicators for the diagnosis of AC.

SECONDARY OUTCOMES:
Heart rate variability assessment | Measured immediately after intervention.
  Dynamic electrocardiogram recording analysis of sympathetic vagal activity.
Neurotransmitter detection analysis | Measured immediately after intervention.
  Serum ACh, NO and VIP

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, China

REFERENCES:
- [Background] Pomenti S, Blackett JW, Jodorkovsky D. Achalasia: Diagnosis, Management and Surveillance. Gastroenterol Clin North Am. 2021 Dec;50(4):721-736. doi: 10.1016/j.gtc.2021.07.001. Epub 2021 Oct 2. PMID 34717867
- [Background] Schlottmann F, Patti MG. Esophageal achalasia: current diagnosis and treatment. Expert Rev Gastroenterol Hepatol. 2018 Jul;12(7):711-721. doi: 10.1080/17474124.2018.1481748. Epub 2018 Jun 8. PMID 29804476
- [Background] Mari A, Abu Baker F, Pellicano R, Khoury T. Diagnosis and Management of Achalasia: Updates of the Last Two Years. J Clin Med. 2021 Aug 16;10(16):3607. doi: 10.3390/jcm10163607. PMID 34441901
- [Background] Gregersen H, Lo KM. Pathophysiology and treatment of achalasia in a muscle mechanical perspective. Ann N Y Acad Sci. 2018 Dec;1434(1):173-184. doi: 10.1111/nyas.13711. Epub 2018 May 14. PMID 29756656
- [Background] Shiwaku H, Sato H, Shimamura Y, Abe H, Shiota J, Sato C, Ominami M, Sakae H, Hata Y, Fukuda H, Ogawa R, Nakamura J, Tatsuta T, Ikebuchi Y, Yokomichi H, Hasegawa S, Inoue H. Risk factors and long-term course of gastroesophageal reflux disease after peroral endoscopic myotomy: A large-scale multicenter cohort study in Japan. Endoscopy. 2022 Sep;54(9):839-847. doi: 10.1055/a-1753-9801. Epub 2022 Feb 16. PMID 35172368
- [Background] Schlottmann F, Neto RML, Herbella FAM, Patti MG. Esophageal Achalasia: Pathophysiology, Clinical Presentation, and Diagnostic Evaluation. Am Surg. 2018 Apr 1;84(4):467-472. PMID 29712590
- [Background] Goyal RK, Padmanabhan R, Sang Q. Neural circuits in swallowing and abdominal vagal afferent-mediated lower esophageal sphincter relaxation. Am J Med. 2001 Dec 3;111 Suppl 8A:95S-105S. doi: 10.1016/s0002-9343(01)00863-4. PMID 11749933
- [Background] Clyburn C, Travagli RA, Browning KN. Acute high-fat diet upregulates glutamatergic signaling in the dorsal motor nucleus of the vagus. Am J Physiol Gastrointest Liver Physiol. 2018 May 1;314(5):G623-G634. doi: 10.1152/ajpgi.00395.2017. Epub 2018 Jan 25. PMID 29368945
- [Background] Browning KN, Carson KE. Central Neurocircuits Regulating Food Intake in Response to Gut Inputs-Preclinical Evidence. Nutrients. 2021 Mar 11;13(3):908. doi: 10.3390/nu13030908. PMID 33799575
- [Background] Farre R, Sifrim D. Regulation of basal tone, relaxation and contraction of the lower oesophageal sphincter. Relevance to drug discovery for oesophageal disorders. Br J Pharmacol. 2008 Mar;153(5):858-69. doi: 10.1038/sj.bjp.0707572. Epub 2007 Nov 12. PMID 17994108
- [Background] Hornby PJ, Abrahams TP. Central control of lower esophageal sphincter relaxation. Am J Med. 2000 Mar 6;108 Suppl 4a:90S-98S. doi: 10.1016/s0002-9343(99)00345-9. PMID 10718459
- [Background] Abrahams TP, Partosoedarso ER, Hornby PJ. Lower oesophageal sphincter relaxation evoked by stimulation of the dorsal motor nucleus of the vagus in ferrets. Neurogastroenterol Motil. 2002 Jun;14(3):295-304. doi: 10.1046/j.1365-2982.2002.00329.x. PMID 12061915
- [Background] Urban DJ, Roth BL. DREADDs (designer receptors exclusively activated by designer drugs): chemogenetic tools with therapeutic utility. Annu Rev Pharmacol Toxicol. 2015;55:399-417. doi: 10.1146/annurev-pharmtox-010814-124803. Epub 2014 Sep 25. PMID 25292433
- [Background] Roth BL. DREADDs for Neuroscientists. Neuron. 2016 Feb 17;89(4):683-94. doi: 10.1016/j.neuron.2016.01.040. PMID 26889809
- [Background] Magnus CJ, Lee PH, Bonaventura J, Zemla R, Gomez JL, Ramirez MH, Hu X, Galvan A, Basu J, Michaelides M, Sternson SM. Ultrapotent chemogenetics for research and potential clinical applications. Science. 2019 Apr 12;364(6436):eaav5282. doi: 10.1126/science.aav5282. Epub 2019 Mar 14. PMID 30872534
- [Background] Nagai Y, Miyakawa N, Takuwa H, Hori Y, Oyama K, Ji B, Takahashi M, Huang XP, Slocum ST, DiBerto JF, Xiong Y, Urushihata T, Hirabayashi T, Fujimoto A, Mimura K, English JG, Liu J, Inoue KI, Kumata K, Seki C, Ono M, Shimojo M, Zhang MR, Tomita Y, Nakahara J, Suhara T, Takada M, Higuchi M, Jin J, Roth BL, Minamimoto T. Deschloroclozapine, a potent and selective chemogenetic actuator enables rapid neuronal and behavioral modulations in mice and monkeys. Nat Neurosci. 2020 Sep;23(9):1157-1167. doi: 10.1038/s41593-020-0661-3. Epub 2020 Jul 6. PMID 32632286
- [Background] Travagli RA, Anselmi L. Vagal neurocircuitry and its influence on gastric motility. Nat Rev Gastroenterol Hepatol. 2016 Jul;13(7):389-401. doi: 10.1038/nrgastro.2016.76. Epub 2016 May 25. PMID 27251213
- [Background] Li J, Xu K, Guo Y, Chen X, Li G, Qi L, Che X. Case evidence of repetitive transcranial magnetic stimulation in the management of refractory irritable bowel syndrome with comorbid depression. Brain Stimul. 2022 Mar-Apr;15(2):434-436. doi: 10.1016/j.brs.2022.01.020. Epub 2022 Feb 11. No abstract available. PMID 35158109
- [Background] Algladi T, Harris M, Whorwell PJ, Paine P, Hamdy S. Modulation of human visceral sensitivity by noninvasive magnetoelectrical neural stimulation in health and irritable bowel syndrome. Pain. 2015 Jul;156(7):1348-1356. doi: 10.1097/j.pain.0000000000000187. PMID 25867123